CLINICAL TRIAL: NCT00752505
Title: A Phase 2 Randomized Double-Blind Placebo-Controlled Crossover Study Assessing The Ability Of Esreboxetine (PNU-165442g) To Improve Cognitive Function In Fibromyalgia Patients.
Brief Title: A Study To Assess Esreboxetine's Effect On Concentration, Memory, Decision Making And Problem Solving In Patients With Fibromyalgia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6061061
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — esreboxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Esreboxetine
- B (Experimental)
  Interventions: Drug: Esreboxetine

INTERVENTIONS:
Drug: Esreboxetine — Tablet once daily either placebo, 4mg or 8mg per day. Subjects will be on active treatment for 4 weeks out of a total of 11 weeks in a crossover dosing
  Arms: A
Drug: Esreboxetine — Tablet once daily either placebo, 4mg or 8mg per day. Subjects will be on active treatment for 4 weeks out of a total of 11 weeks in a crossover dosing
  Arms: B

SUMMARY:
The study is designed to assess if esreboxetine can improve the cognitive function of patients with fibromyalgia. Cognitive function is defined as the ability to concentrate, remember things and make decisions or problem solve. The study is also designed to assess if there is a difference in cognitive function between fibromyalgia patients and matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a recognised diagnosis of fibromyalgia, with defined minimum pain criteria. Control subjects must not have a fibromyalgia diagnosis or symptoms and must match fibromyalgia subjects for age, length of education and gender

Exclusion Criteria:

* Other confounding pain, cognitive disease or impairment, disease that could put the subject at risk or subjects who are on prohibited medications that cannot be washed out.
* Any subjects with a diagnosis of certain psychiatric disorders in particular major depression or suicidal risk. Matched control subjects have similar exclusions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Computer based psychometric tests | 11 week

SECONDARY OUTCOMES:
A questionnaire to evaluate the subjects cognitive status | Once at randomisatoin
A questionnaire to assess the subjects mood | 11 weeks
A question to assess the subjects pain at visits | 11 weeks
A daily diary to assess the subjects pain | 11 weeks
A questionnaire to evaluate the impact the subject perceives fibromyalgia has on their cognitive ability | Once at randomisation
Two questionnaires to assess change in the subjects cognitive ability | 11 weeks
Safety evaluations: medical history, physical and neurological exam, heart rate and blood pressure lying and standing, laboratory tests, electrical heart trace (ECG), adverse event collection, assessment of suicidal risk | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Fort Walton Beach, Florida
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061061&StudyName=A%20Phase%202%20Randomized%20Double-Blind%20Placebo-Controlled%20Crossover%20Study%20Assessing%20The%20Ability%20Of%20Esreboxetine%20%28PNU-165442g%29%20To%20Improve%20Cognitive%20Function%20In%20Fibromyalgia%20Patients